CLINICAL TRIAL: NCT00530738
Title: Efficacy, Safety and Quality of Life of a Long-term Home Parenteral Nutrition Regimen With Either LIPIDEM® or LIPOFUNDIN® MCT a Mono-center, Randomized, Double Blind Study
Brief Title: Safety and Efficacy of Longterm HPN With Two Lipid Emulsions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HC-G-H-0503; EudraCT-Nr.: 2005-001938-32
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Malnutrition
Keywords: HPN; lipid emulsion; long term; insufficient enteral resorption capacity
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): treatment with Lipoplus & Nutriflex plus (commercially available and marketed 2 Chamber Bag)
  Interventions: Drug: Lipoplus
- 2 (Active Comparator): treatment with Lipofundin MCT & Nutriflex plus (commercially available and marketed 2 Chamber Bag)
  Interventions: Drug: Lipofundin MCT

INTERVENTIONS:
Drug: Lipoplus — i.v. fat emulsion for parenteral nutrition
  Arms: 1
Drug: Lipofundin MCT — i.V. fat emulsion for parenteral nutrition
  Arms: 2

SUMMARY:
It is the purpose of this trial to provide evidence for safety and efficacy of long term home parenteral nutrition with either Lipofundin MCT or Lipoplus in patients with proven insufficient enteral resorption.

DETAILED DESCRIPTION:
Long term parenteral nutrition is indicated in the home care setting of patients who are unable to completely cover their daily caloric requirements by oral/enteral nutrition due to e.g. pre existing malnutrition or compromised intestinal absorption.

An appropriate nutritional supplementation ensuring the provision of patients basic requirement of amino acids, glucose, lipids, micronutrients and electrolytes is therefore required to stop weight loss, increase quality of life and to reduce unfavorable consequences of malnutrition in those patients.

Major causes for malnutrition and compromised intestinal absorption are malignant processes. Tumor cachexia, weight loss due to insufficient nutrition of < 60 -80 % of the calculated substrate need for > 14 days, antineoplastic therapy and surgical intervention are consequences of the malignant disease and lead to catabolic processes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age: 18-80 years
* Male and female patients
* Patients with a newly indicated need of long-term home parenteral nutrition (HPN) for at least 8 weeks
* Patients with an insufficient resorption capacity of the colon that may not be compensated by enteral nutrition
* mentally and physically able to adhere to study procedures.
* Females agree to apply adequate contraception

Exclusion Criteria:

* Participation in a clinical study with an investigational drug within one month prior to the start of study
* Patients with sepsis, severe sepsis and septic shock
* Known or suspected drug abuse
* General contra indications for infusion therapy such as acute pulmonary edema, hyperhydration and decompensated cardiac insufficiency
* Pregnancy and lactation
* Autoimmune disease as e.g. HIV
* Known hypersensitivity to egg-, soy-, and fish proteins or any of the ingredients
* Hemodynamic failure of any origin (hemorrhagic shock, myocardial infarction, cardiac failure)
* Alterations of coagulation (thrombocytes <150.000 mm3), PT < 50%, PTT > 40 sec
* Diabetes mellitus with known ketoacidosis within 7 days before onset of study
* Renal insufficiency with serum creatinine > 1.4 mg/dL(>124 mmol/L)
* Patients with severe liver dysfunction with bilirubin >2.5 mg/dL (> 43 µmol/L)
* Lipid disorders, in particular fasting serum triglycerides > 250 mg/dL (>2.86 mmol/L)
* necrotizing pancreatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Proof of non-inferiority of a HPN regimen containing Lipidem compared to a Lipofundin MCT containing regimen as indicated by the BMI | 8 weeks

SECONDARY OUTCOMES:
Evaluation of beneficial effects of a long-term HPN-regimen with Lipidem on Quality of Life and body composition | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Thul, MD, Principal Investigator — Charité, University Hospital Berlin
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Derived] Bohnert H, Maurer M, Calder PC, Pratschke J, Thul P, Muller V. Efficacy of a long-term home parenteral nutrition regimen containing fish oil-derived n-3 polyunsaturated fatty acids: a single-centre, randomized, double blind study. Nutr J. 2018 Nov 30;17(1):113. doi: 10.1186/s12937-018-0419-x. PMID 30501620